CLINICAL TRIAL: NCT04810988
Title: Variable-dose Support in an Online Mental Health Intervention
Brief Title: Outcomes of a Self-guided Versus Therapist-guided Online Mental Health Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: Charles Lafitte Foundation (Unknown)
Responsible Party: Principal Investigator, Heather Parnell, PhD Candidate, Duke University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2021-0292
Record Dates: First submitted 2021-03-18; First posted 2021-03-23 (Actual); Last update posted 2024-07-22 (Actual); Status verified 2024-07

CONDITIONS: Depression; Anxiety; Mood
Keywords: depression; anxiety; mood; mood disorder; digital health; mHealth; unified protocol; pilot study
MeSH Terms: conditions — Depression; Anxiety Disorders; Mood Disorders | interventions — Cor a I protein, hazel

STUDY DESIGN:
Intervention Model Description: Eligible, consented participants will be immediately randomized to one of two arms and remain in that arm for the duration of the study.
Masking Description: Neither participants nor study therapists will be blinded to participant condition, as it is not feasible to blind to whether or not someone is receiving therapist support.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Unsupported (Active Comparator): Participants in this arm will receive a 12-week Unified Protocol intervention delivered via the same web platform. Each week, participants will complete the following content:
  1. depression survey,
  2. anxiety survey,
  3. information about their symptom change over time,
  4. psychoeducational text
  5. practice exercises,
  6. home practice instructions,
  7. writing exercise,
  8. home practice worksheets.
  In the first week, participants will receive an emailed welcome message followed by a link to the first week's content. For every following week, participants will receive an email at the start of the week with automatically generated feedback on intervention usage, behavior change, and symptom change, as well as the link to the new week's intervention content.
  Interventions: Behavioral: Unified Protocol
- Partially Supported (Experimental): Participants in the partially supported arm will receive all aspects of the intervention described above, with no differences between arms for the first seven weeks of the intervention (Modules 1-6). Participants will be introduced to their study therapist in week 8, at the start of Module 7 via email. During Module 7 (exposure; weeks 8-11), participants will receive four video therapy sessions. Session content will be based on principles of exposure therapy (developing a personalized exposure hierarchy, live demonstrations of exposure exercises, in-session exposure practices, post-exposure processing, home practice assignments, and therapist feedback).
  Interventions: Behavioral: Unified Protocol; Behavioral: Therapist Support

INTERVENTIONS:
Behavioral: Unified Protocol — The Unified Protocol is an empirically supported, transdiagnostic treatment for emotion disorders based on principles of cognitive behavioral therapy. Treatment focuses on increasing awareness of maladaptive thoughts and behaviors and decreasing avoidance of emotions and physiological sensations. Module 1 is focused on increasing motivation, readiness and self-efficacy for change. Module 2 focuses on increasing understanding and awareness of emotions. Module 3 is focused on further expanding awareness of emotions. Module 4 focuses on the role of thoughts in emotional disorders. Module 5 is focused on the role of behaviors in emotional disorders. Module 6 focuses on the role of physical sensations in emotional disorders. Module 7 focuses on exposure to interoceptive and situational triggers for emotions. Module 8 is focused on maintenance of treatment progress and relapse prevention.
  Other Names: Hazel
Behavioral: Therapist Support — 4 video calls with study therapists
  Arms: Partially Supported

SUMMARY:
This is a pilot study of an online mental health treatment. The goals of the study are to determine the feasibility of an online treatment for depression and anxiety symptoms with little-to-no human support, in a sample of 50 adults with limited educational attainment. The treatment is based on the Unified Protocol, an evidence-based treatment for mood and anxiety symptoms. The study will enroll participants on a rolling basis until reaching the goal of 50 participants. The intervention lasts 16 weeks, with 12 weeks of online treatment focused on increasing mindfulness, decreasing avoidance, and increasing cognitive flexibility in order to decrease depression and anxiety symptoms. Participants will complete surveys about their symptoms and how they feel about the treatment to help us establish the feasibility of a larger trial.

DETAILED DESCRIPTION:
The study is a 12-week, randomized controlled trial ("Hazel") comparing an intervention for depression and anxiety symptoms with two different levels of support. Eligible participants will be randomized to receive: 1) a Unified Protocol intervention with 4 weeks of human support during exposure exercises in weeks 8-11 ("Partially Supported"); or 2) a Unified Protocol intervention without support at any point (the "Unsupported" arm). At 4 weeks post-intervention, participants will be sent a link to complete follow-up survey measures for depression and anxiety symptoms.

The Unified Protocol is an empirically supported, transdiagnostic treatment for emotion disorders based on principles of cognitive behavioral therapy.27 The Unified Protocol can be delivered in 12 to 18 weeks, with one one-hour session per week. Treatment focuses on increasing awareness of maladaptive thoughts and behaviors while decreasing avoidance of emotions and physiological sensations. Each week, patients receive psychoeducation, complete in-session practice exercises and self-monitor symptom change. At the end of each session, patients are assigned a home practice assignment to increase adaptive coping and generalize skill use outside of the therapy room.

Participants in both arms will receive a 12-week Unified Protocol intervention delivered via the same web platform (REDCap). The intervention will include all 8 modules of the Unified Protocol. Every week, participants will be directed to complete the following content:

1. depression symptom survey,
2. anxiety symptom survey,
3. information about their symptom change over time,
4. psychoeducational text
5. practice exercises,
6. home practice instructions,
7. writing exercise, and
8. home practice worksheet(s).

The symptom surveys, symptom graph and writing exercise will remain the same each week. The psychoeducational text, practice exercises and homework assignments will vary based on that week's topic. For the writing exercise, participants will be prompted to write notes on their take-aways, questions about the material, and ways they can incorporate the lesson into their upcoming week. The investigators will aim to write as much text as possible at a 5th grade reading level, based on evidence that 52% of US residents read English at a 5th-grade level or below.

Participants randomized to the unsupported arm will receive the intervention exactly as described above, with no additional components. Completion of all weeks will be entirely self- guided, to emulate a publicly available, standalone intervention.

Participants randomized to the partially supported arm will receive all aspects of the intervention described above, with no differences between arms for the first seven weeks of the intervention (Modules 1-6). Participants in this arm will be introduced to their assigned study therapist in week 8, at the start of Module 7 via email. During Module 7 (exposure; weeks 8-11), participants in this arm will receive four video therapy sessions. These sessions will entail synchronous, video-call contact with their assigned study therapist, and session content will be based on principles of exposure therapy. The first session will entail developing a personalized exposure hierarchy, which will inform subsequent in-session and home practice assignments. In all sessions, study therapists will do live demonstrations of exposure exercises, monitor participants during exposure practice and provide feedback as clinically indicated, guide participants through post-exposure processing, and assign in-vivo exposure practices for homework. In the second through fourth sessions, study therapists will also review and provide feedback on participants' home practice.

Study therapists will be clinical psychology graduate students at Duke University and will be trained and supervised by Dr. Clair Robbins, a clinical associate at Duke and expert in the Unified Protocol. Dr. Robbins is expected to pass licensure exams during the Spring 2021 semester. Until then, umbrella supervision will be provided by Dr. M. Zach Rosenthal, a North Carolina-license psychologist and director of Duke's Cognitive Behavioral Research and Treatment Program.

On recruitment and participant materials, the study will be referred to by the name "Hazel." Hazel was chosen as a name because it is a relatively uncommon word that is both a name and a noun. The investigators' hope is that using a study title that can be a name will evoke a sense of warmth and personalization in the online intervention. At the same time, "Hazel" is not exclusively used a name, which the investigators hope will prevent undue confusion or misleading respondents into thinking Hazel is a human therapist. Finally, the investigators hope that its relatively uncommon usage will help prevent confusion with any other similar studies or programs. The name Hazel is incorporated into study materials in terms of color scheme and logo. At the end of the intervention, the hazelnut logo used throughout Hazel will be transformed into a hazelnut tree sprout, symbolizing both the ways participants have grown over the course of the intervention and the possibility for ongoing growth as they continue applying their new skills after the intervention period ends.

ELIGIBILITY:
Inclusion Criteria:

* 18+ years old
* Fluent in reading and writing English
* Internet/data plan and computer/tablet/phone access for length of study
* Overall Depression Severity and Impairment Scale (ODSIS) and/or Overall Anxiety Severity and Impairment Scale (OASIS) summary score >= 8
* Live in North Carolina for the duration of the study

Exclusion Criteria:

* Educational attainment greater than high school diploma/equivalent
* Currently receiving other psychotherapy or planning to receive other psychotherapy during course of intervention
* >=8 sessions of cognitive-behavioral therapy in past 12 months
* Currently taking psychiatric medications or planning to take psychiatric medications during course of intervention
* Current suicidality, operationalized as a positive result on the Ask Suicide-Screening Questions (ASQ) Tool
* Self-harm in past 12 months
* Current psychosis, as measured by Mini International Neuropsychiatric Interview Subsection K. Psychotic Disorders
* Substance abuse (other than nicotine, cannabis or caffeine) in the past 12 months, as measured by Structured Clinical Interview for The Diagnostic and Statistical Manual of Mental Disorders-5 substance use disorders subsection (past 12 months only)
* BMI <= 18.5

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2021-04-07 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
Change Between Baseline and Post-Treatment System Usability Scale Score | through study completion, an average of 12 weeks
  10-item, validated self-report user experience survey for digital systems answered on a five-point Likert scale
Weekly Change in Willingness to Refer | through study completion, an average of 12 weeks
  yes/no question if participants would recommend the intervention to others
Total Number of Referrals (Sum Score) | through study completion, an average of 12 weeks
  pts who select yes for willingness to refer will be given option to actually make referrals. this will calculate a sum score of total number of referrals
Change in Cognitive Flexibility Inventory Score | through study completion, an average of 12 weeks
  20-item measure of cognitive flexibility designed to be used for repeated measures over the course of an intervention
Change in Cognitive and Affective Mindfulness Scale-Revised Score | through study completion, an average of 12 weeks
  10-item questionnaire that assesses mindfulness of thoughts and emotions
Change in COPE Inventory - Avoidance Factor Score | through study completion, an average of 12 weeks
  COPE Inventory is a survey of coping strategies with 60-items split across 15 4-item scales; factor analysis has identified a 16-item avoidance factor, comprising 4 4-item subscales (mental disengagement, denial, behavioral disengagement, and substance use) which will be used for this study as the remaining items on the full COPE Inventory are not related to primary mechanisms of change in this intervention

SECONDARY OUTCOMES:
Change in Overall Depression Severity and Impairment Scale Score | through study completion, an average of 12 weeks
  A 5-question survey measure of depression symptoms
Change in Overall Anxiety Severity and Impairment Scale Score | through study completion, an average of 12 weeks
  A 5-question survey measure of anxiety symptoms

CONTACTS AND LOCATIONS:
Overall Officials: Jack Brooks, MA, Study Director — Duke University; Gary G Bennett, PhD, Principal Investigator — Duke University
Locations (1):
- Duke University, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No
There is no plan to share IPD with researchers other than those directly involved with the study and on the study Institutional Review Board.